CLINICAL TRIAL: NCT04237831
Title: A Phase 1, Open-Label, Multiple-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BMS-986259 in Participants With Varying Degrees of Renal Function
Brief Title: A Study to Evaluate the Pharmacokinetics (Drug Levels and Metabolism), Safety, and Tolerability of BMS-986259 in Participants With Various Levels of Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CV019-008
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Normal Renal Function (Experimental)
  Interventions: Drug: BMS-986259
- Arm B: Mild Renal Impairment (Experimental)
  Interventions: Drug: BMS-986259
- Arm C: Moderate Renal Impairment (Experimental)
  Interventions: Drug: BMS-986259
- Arm D: Severe Renal Impairment (Experimental)
  Interventions: Drug: BMS-986259

INTERVENTIONS:
Drug: BMS-986259 — Specified Dose on Specified Days

SUMMARY:
A study to evaluate the drug effect, safety, and tolerability of BMS-986259 in participants with different levels of kidney function

DETAILED DESCRIPTION:
Recruitment temporarily on hold due to COVID-19

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Participant must have renal impairment, as defined by eGFR at screening using the Chronic Kidney Disease Epidemiology (CKD-EPI) equation
* No change in medications to control Chronic Kidney Disease (CKD) for at least 2 weeks prior to dosing, and if possible, during confinement in the clinical research unit (CRU), except those cleared by the investigator and Medical Monitor.
* Participants with normal renal function at screening, based upon the opinion of the investigator's medical evaluation.
* Medically well-controlled disorders (eg, stable chronic asthma, allergy) are permitted if the treatment for the disease does not interfere with the study.
* Women and men must use highly effective methods of contraception for the duration of treatment

Exclusion Criteria:

* History of any significant drug allergy or drug-related Serious Adverse Events (SAE) (such as anaphylaxis or hepatotoxicity)
* Positive results for drugs abuse in urine/saliva
* Participants undergoing any method of dialysis (eg, hemodialysis, peritoneal dialysis) within the last 3 months or with anticipated need for dialysis during the study
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory assessments beyond what is consistent with the target population
* Known previous exposure to BMS-986259

Other inclusion/exclusion criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Maximum plasma Concentration (Cmax) of BMS-986259 in Blood serum | Day 1 and Day 8
Time to reach maximum concentration in plasma (Tmax) of BMS-986259 in blood serum | Day 1 and Day 8
Area under the concentration- time curve over the dosing interval of BMS-986259 in blood serum - AUC(TAU) | Day 1 and Day 8
Concentration of BMS-986259 in blood serum at 24 hours (C24) | Day 1 and Day 8
Area under the concentration-time curve of BMS-986259 from time 0 (dosing) to the time of the last quantifiable - AUC(0-T) | Day 8
Accumulation ratio in the maximum plasma concentration of BMS-986259 in blood serum -AR(Cmax) | Day 8
Accumulation ratio of Area under the concentration-time curve in BMS-986259 over the dosing interval -AR (AUC [TAU]) | Day 8
Accumulation ratio concentration of BMS-986259 at 24 hours- AR(C24) | Day 8
Terminal elimination half-life of BMS-986259 (T-HALF) | Day 8
Apparent total clearance of BMS-986259 at steady-state (CLss/F) | Day 8
Apparent volume of distribution of BMS-986259 at terminal phase at steady-state (Vss/F) | Day 8

SECONDARY OUTCOMES:
Incidence of Non serious Adverse Events (AEs) | Up to 4 months
Incidence of Serious Adverse Events (SAEs) | Up to 4 months
Incidence of AEs leading to discontinuation | Up to 4 months
Number of clinically significant changes in vital signs | Up to 4 months
Number in clinically significant changes in Electrocardiogram (ECG) | Up to 4 months
Number of clinically significant changes in physical examinations | Up to 4 months
Number of clinically significant changes in clinical laboratory tests | Up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Prism Clinical Research, Saint Paul, Minnesota

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm